CLINICAL TRIAL: NCT05296928
Title: The Effect of the Umbilicus and Sub-umbilicus Incisions Used in Laparoscopic Gynecological Surgeries on the Postoperative Pain Score
Brief Title: Postoperative Pain Score of Laparoscopic Gynecological Surgeries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baskent University (Other)
Responsible Party: Principal Investigator, Didem Alkaş Yağınç, Principal Investigator, Baskent University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: BaskentU KA21/186
Record Dates: First submitted 2021-10-28; First posted 2022-03-25 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Surgical Incision; Gynecologic Surgery; Postoperative Pain
Keywords: laparoscopic surgery; umbilical incision; postoperative pain score
MeSH Terms: conditions — Surgical Wound; Pain, Postoperative

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- umbilical incision (Experimental): Placing the laparoscopic trocar by cutting the umbilicus directly at the entrance to the abdomen
  Interventions: Procedure: laparoscopic incision
- subumbilical incision (Active Comparator): Placing a laparoscopic trocar by making a sub-umbilicus incision at the entrance to the abdomen
  Interventions: Procedure: laparoscopic incision

INTERVENTIONS:
Procedure: laparoscopic incision — laparoscopic umbilical trocar entry pathways

SUMMARY:
In this study, it was aimed to compare the embryonic route, the umbilicus, and the sub-umbilicus incision in terms of postoperative pain scoring. For this purpose, in laparoscopic hysterectomies performed for benign reasons, it is planned to measure the pain score at the 8th hour and 1st day postoperatively in the umbilicus and subumbilical incision. Visual analog scoring system will be used for pain scoring.

DETAILED DESCRIPTION:
In this prospective randomized study, Baskent University Adana Dr. Turgut Noyan Application and Research Center for benign reasons (myomas that cause abnormal uterine bleeding, resistant to medical and hysterescopic surgery, treatment-resistant adenomyosis in which the uterus reaches 12 weeks of gestation, recurrent endometrial hyperplasia, endometriosis, stage 1 endometrial cancers that only underwent hysterectomy) in laparoscopic hysterectomies; at the entrance to the abdomen, it is planned to apply the umbilicus, which is the anatomical route, to some of the patients, and to the other part of the sub-umbilicus incision. It will be compared in terms of pain score on the 8th hour and 1st day after surgery. The minimum quorum for each group was determined by calculating 41 and taking a total of 82 patients. The simple randomization technique will be applied in the distribution to the study sets. Based on the studies, it is thought that the anatomical path may be less painful.

ELIGIBILITY:
Inclusion Criteria

1. Patients who underwent laparoscopic hysterectomy for benign reasons
2. Stage 1 endometrial cancers that only underwent hysterectomy

Exclusion Criteria:

1. Malign disorders
2. Uterus larger than 12 weeks of gestation

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2022-07-07 (Actual); Primary Completion 2023-04-27 (Actual); Study Completion 2023-05-27 (Actual)

PRIMARY OUTCOMES:
postoperative pain score | 8 hour
  The umbilicus, which is the embryonic pathway used in laparoscopic surgery, is expected to cause less postoperative pain.In the Visual Analog Score to be used as the pain measurement criterion, '0' indicates no pain, while '10' defines the most severe pain.

SECONDARY OUTCOMES:
postoperative pain score after 24 hour | 24 hour
  The umbilicus, which is the embryonic pathway used in laparoscopic surgery, is expected to cause less postoperative pain.In the Visual Analog Score to be used as the pain measurement criterion, '0' indicates no pain, while '10' defines the most severe pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Başkent University Adana Dr. Turgut Noyan Application and Research Center, Adana, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No